CLINICAL TRIAL: NCT04323059
Title: Effectiveness, Tolerability and Safety of Standardized Milk-based, Standardized Non-milk Based and Hospital-based Formulations in the Management of Moderate Acute Malnutrition in Underfive Children: A Randomized Clinical Trial
Brief Title: Effectiveness, Tolerability and Safety of Three Formulations in Underfives With Moderate Acute Malnutrition
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Ekong E. Udoh (Other)
Responsible Party: Sponsor-Investigator, Dr. Ekong E. Udoh, DOCTOR, University of Uyo Teaching Hospital
Organization: University of Uyo Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UUTH/AD/S/96/VOL.XXI/341
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Malnutrition; Moderate
Keywords: Nutrition; Formulations; Moderate; Malnutrition; Underfives
MeSH Terms: conditions — Malnutrition; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: The study participants will be randomized into three different intervention groups. Based on the group of assignment, the participants will receive either the standardized milk-based formulation, the standardized non-milk based formulation or the hospital-based formulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized milk-based formulation (Experimental): Formulation of maize with milk that is rich in methionine
  Interventions: Dietary Supplement: Standardized milk-based formulation
- Standardized non-milk based formulation (Experimental): Formulation of maize with soybeans that is rich in methionine and lysine
  Interventions: Dietary Supplement: Standardized milk-based formulation
- Hospital-based formulation (Active Comparator): Formulation of maize, milk and soybeans
  Interventions: Dietary Supplement: Standardized milk-based formulation

INTERVENTIONS:
Dietary Supplement: Standardized milk-based formulation — Nutritional formulations prepared from locally available food stuffs for reversing childhood malnutrition
  Other Names: Standardized non-milk based formulation; Hospital-based formulation

SUMMARY:
This is a randomized clinical trial aimed at evaluating the effectiveness, tolerability and safety of standardized milk-based formulation, standardized non-milk based formulation and a hospital-based formulation in the management of children aged 6 - 59 months with moderate acute malnutrition. Eligible children will be randomized into one of the three intervention arms and given supplementary doses of the formulations at 50% of their daily caloric requirement for a period of four months based on the group of their assignment. The remainder will be obtained from their regular family diets. The clinical features, anthropometric measurements and laboratory parameters of the children will be assessed at baseline. The children will be followed up on two weekly basis for a period of four months during which further clinical assessment, anthropometric measurements and laboratory evaluations will be performed. The outcome measures will be determined based on "per protocol analysis".

DETAILED DESCRIPTION:
Childhood malnutrition is presently a leading cause of underfive morbidity and mortality globally. The impact of the condition is most severe in the first 1000 days of life with resultant impairment in physical, neurologic, immunologic and metabolic development.

Undernutrition, the commoner form of childhood malnutrition, is usually classified as underweight (weight-for-age Z score < -2), stunting (height-for-age Z score <-2), wasting (weight-for-height Z score < -2) or edematous malnutrition (kwashiorkor) in relation to the World Health Organization standard reference values for age and sex. It is further sub-classified into severe acute malnutrition (SAM) wherein z score is <-3 and moderate acute malnutrition (MAM) wherein z score is between -2 and -3.(1) MAM accounts for about 70.0% of all malnutrition-related childhood deaths.

Children with MAM are currently managed using community-based approach. This approach entails early detection and treatment of children with MAM in the community, timely referral to inpatient care for those that progress to SAM or develop complications, and subsequent follow up in the community at discharge. MAM is usually managed by nutrition education of the caregivers on preparation of nutritious, palatable and culturally acceptable food from locally available food stuffs like banana porridge or corn gruel fortified with legume (mashed groundnut or soya bean), crayfish, palm oil, powdered milk and vegetables. The second strategy is by Ready-to-use therapeutic foods (RUTFs). (2) The main drawback of the RUTFs is that they are usually provided by external donor agencies and as such, not always available in settings where childhood malnutrition is endemic. Children treated with RUTFs are therefore at risk of progressing to SAM or dying when the formulations are no longer available. There is currently no consensus on the appropriate nutritional formulation for community-based management of MAM in children in endemic regions. It is therefore imperative to evaluate the effect of readily available formulations that are comparable to the RUTFs in community-based management of childhood MAM in endemic regions. (3) The standardized milk-based formulation (SMBF), the standardized non milk-based formulation (SNMBF) and the hospital-based formulation (HBF) are examples of formulations that are readily available in the country. The SMBF consists of maize and is rich in methionine, the SNMBF consists of maize and soybeans, and is rich in methionine and lysine while the HBF consist of a combination of maize, milk and soybeans. The nutrient composition of the above-mentioned formulations is similar to that of the RUTFs, making them suitable for community-based management of MAM. However, no clinical trial has so far been conducted to evaluate their effect in managing underfive children with MAM. The cost effectiveness of the various formulations will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6 - 59 months with moderate acute malnutrition (weight-for-height between -2 and -3 Z scores or mid upper arm circumference of 11.5 cm - 12.5 cm).
2. Children whose parents/guardian consent to their participation and agree to bring the children/wards to the health facility throughout the period of the study.

Exclusion Criteria:

1. Children with chronic illnesses that may affect growth {(cardiac disease, renal disease, tuberculosis (chronic cough, history of contact with an adult with chronic cough, poor growth, chest infection not responding to antibiotics) liver disease, HIV/AIDS}
2. Children with feeding difficulties eg. Gastroesophageal reflux diseases, cleft palate
3. Children with diarrhoea
4. Children with neurological diseases eg. Cerebral palsy
5. Children less than 6 months or more 59 months of age

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
weight-for-height | Four months
  Improvement in weight-for-height at two weekly intervals

SECONDARY OUTCOMES:
Recovery from moderate acute malnutrition | Four month
  Proportion of children whose weight-for-height z score improved from <-2 to ≥ 2
Adverse events | Four months
  The number of children that develop and undesirable gastrointestinal or extraintestinal disorder

CONTACTS AND LOCATIONS:
Overall Officials: Ekong E Udoh, FWACPaed, Principal Investigator — University of Uyo Teaching Hospital, Uyo, Akwa Ibom State, Nigeria; Sunday B Adesina, FWACPaed, Study Director — University of Uyo Teaching Hospital, Uyo, Akwa Ibom State, Nigeria; Blessing N Nwazuluoke, BSc, Study Chair — University of Uyo Teaching Hospital, Uyo, Akwa Ibom State, Nigeria
Locations (3):
- Nigeria (3):
  - Primary Health Centre, Okpoediuse, Ibiono Ibom, Akwa Ibom State
  - Primary Health Centre, Adadiah, Uruan, Akwa Ibom State
  - Primary Health centre, Mbak-Etoi, Uyo, Akwa Ibom State

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available to other researchers by the Principal Investigator on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available for two years after completion of the trial
Access Criteria: Any investigator that request for it within the time frame will be given

REFERENCES:
- [Background] Seetharaman N, Chacko TV, Shankar SLR, Matthew AC. Measuring malnutrition - the roles of Z scores and the composite index of anthropometric failure. Indian Journal of Community Medicine. 2007; 32 (1): 35-39.
- [Background] Vijay DW, Bhawesh RD. Ready to use therapeutic food (RUTF): An overview.. Advances in life Sciences and Health. 2015; 2 (1): 1-15.
- [Background] Choudhury N, Ahmed T, Hossain MI, Islam MM, Sarker SA, Zeilani M, Clemens JD. Ready-to-Use Therapeutic Food Made From Locally Available Food Ingredients Is Well Accepted by Children Having Severe Acute Malnutrition in Bangladesh. Food Nutr Bull. 2018 Mar;39(1):116-126. doi: 10.1177/0379572117743929. Epub 2017 Dec 19. PMID 29258336